CLINICAL TRIAL: NCT05634070
Title: Clinical Trial Evaluating Medical-grade Polycaprolactone-PCL Pectus Scaffold Implantation with Autologous Fat Grafting for Pectus Excavatum Camouflage (IT)
Brief Title: Pectus Excavatum Camouflage (IT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BellaSeno GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-PEC-002
Record Dates: First submitted 2022-11-09; First posted 2022-12-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insertion of a custom-made 3D printed medical-grade polycaprolactone scaffold (Experimental): Insertion of a custom-made 3D printed medical-grade polycaprolactone scaffold in the thorax region with autologous fat graft to camouflage pectus excavatum defect.
  Interventions: Device: PCL Pectus scaffold implantation and autologous fat grafting

INTERVENTIONS:
Device: PCL Pectus scaffold implantation and autologous fat grafting — A suitable incision will be made using a scalpel and diathermy following standard surgical procedures.The implant pocket shall be rinsed with saline. The PCL Pectus Scaffold shall be inserted into the pocket following the Instruction for Use and fixed to the thoracic wall using 2 to 4 sutures. The device shall not be modified for any patient in any manner. The incision shall be closed using 2-0 Vicryl or Monocryl and 3-0 Monocryl sutures, if applicable. Number of layers to be sutured will be decided by the PI for each patient. Sterile bandaging as well as Steri-Strips shall be applied on the sutures. A prophylactic antibiotic such as Cefazolin 1g (3 shots per day x 2 days) shall be administered to the patient. In case the patient has Cefazolin allergy, Clindamycin 600 mg shall be prescribed. Autologous Fat Grafting procedure shall be performed immediately after implantation. The patients shall be hospitalized for the necessary number of days under clinical observation.

SUMMARY:
The clinical study evaluates the use of a custom-made medical-grade polycaprolactone-PCL Pectus scaffold implantation with Autologous Fat Grafting for pectus excavatum camouflage (IT). The study aims to demonstrate the safety and clinical performance of the insertion of an absorbable "medical-grade polycaprolactone-PCL Pectus Scaffold" in the thorax region with Autologous Fat Grafting in the correction of congenital Pectus Excavatum unsuitable for conventional treatment with stable cardio-respiratory function.

The PCL Pectus Scaffold-based design has the potential to induce sustained regeneration to fill large volume pectus excavatum defects, with the added benefit of being light weight and resorbable, thus not affecting the patients function capacity and reducing the risk of implant-related complications.

DETAILED DESCRIPTION:
A 3D printed custom-made scaffold made of medical-grade polycaprolactone (m-PCL) is planned to be implanted to correct pectus excavatum defects.

Participants will be recruited at the Meyer Hospital (Florence, Italy). The patient is assessed clinically by the PI with a direct history and examination, in conjunction with the imaging reviewed by the Principal Investigator and his team. Imaging is organised through the Meyer Hospital imaging department and includes chest CT and MRI. Patients will be formally enrolled into the trial after written informed consent is obtained from the patients and from their parents/legal guardian (in case of minor patients). If the patient is deemed suitable and satisfy the inclusion and exclusion criteria, as assessed by the Principal Investigator and his team, a custom-made scaffold is designed based on his/her medical-imaging.

The procedure for implantation of the scaffold is similar to the procedure for implantation of silicone implants. A small incision is made in the chest, a pre-sternal pocked is defined, following this an empty scaffold is implanted at the site of the defect (pectus excavatum) with skin closed directly over it. At the same intervention, autologous fat transfer is performed, harvesting fat from available donor sites such as the thighs and abdomen - depending on scaffold volume and patient morphology. The scaffold provides structural stability to the infiltration of the tissue inside the scaffold. Once the scaffold is fully absorbed, the tissue, which infiltrated it is expected to provide structural stability to the void defect and potentially ensuring a stable outcome.

After the scaffold implantation and fat grafting procedure, patients will remain an inpatient for the necessary number of days after the surgery. In uncomplicated cases, patients will be reviewed at trial required follow up visits at 1, 3-, 6-, 12- and 24-months post-surgery. Each follow up visit will include routine clinical assessments, review of adverse events and medications, repeat MRI scans and completion of questionnaires for the patients. The focus of these assessments is to identify complications, while establishing clinical and radiological evidence of soft tissue retention.

All appointments and clinical assessment will be documented in the patient medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Genetic female patients of age 14 years and up OR Genetic male patients of age 16 years and up without cardiopulmonary compromise seeking correction or improvement of pectus excavatum-associated with anterior chest wall deformity and/or congenital defect.
2. Patient willing and able to comply with the study requirements (e.g., all scheduled appointments).
3. Patient is eligible to undergo MRI (i.e., no implanted metal or metal devices, no history of severe claustrophobia).
4. Patient and his/her parents/legal guardian (in case of minor patients) capable of providing valid written informed consent.
5. Have sufficient body fat for homologous transplantation.
6. The patient/Guardian has "realistic" expectations of surgical results as determined by the PI.

Exclusion Criteria:

1. Genetic females less than 14 years of age at the time of surgery.
2. Genetic males less than 16 years of age at the time of surgery.
3. Active infection anywhere in the body.
4. Patient chest wall tissue is clinically incompatible for the procedure as determined by PI.
5. Compromised vascularity in the pectoralis muscle and subcutaneous tissue.
6. Patient and is/her parents/legal guardian (in case of minor patients) unwilling or unable to provide fully informed consent including but not limited to patients with intellectual or mental impairment.
7. Patient with a known history of immunodeficiency including HIV, concomitant systemic corticosteroid therapy, chemotherapy, synchronous haematological malignancy, or other cause for secondary/primary immunodeficiency.
8. Known severe concurrent or inter-current illness including cardiovascular, respiratory, or immunological illness, psychiatric disorders, alcohol or chemical dependence, possible allergies that would, in the opinion of the Co-ordinating Principal Investigator, compromise their safety or compliance or interfere with interpretation of study results.
9. Patient with unstable cardiac or respiratory function due to pectus excavatum or those still requiring functional repair.
10. Body mass Index (BMI below 20 and above 30 (patients with a BMI above 30 may still be eligible pending assessment by investigating team and documentation of rationale).
11. Female patients who are currently pregnant or breast feeding, or who are planning to become pregnant within two years after the pectus excavatum camouflage surgery.
12. Female patients of childbearing potential without an appropriate contraceptive method.
13. Patient ineligible to undergo MRI.
14. Patient life expectancy < 36 months.
15. Patient unable or unwilling to comply with the treatment protocol.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events and serious adverse events from the time of surgery to the end of study visit. | Assessed at 24 post-surgery months
  Clinical safety will be assessed by documenting all adverse events regardless of whether they are related to the trial in an adverse events report form - described in detail in the case report form (CRF). These will be carefully evaluated by the principal investigator.
Change in (fat) volume % and soft tissue retention % within the scaffold (radiological and/or clinical) from the time of surgery to the end of study visit using radiological and clinical assessments | Assessed at 1-,6-,12-,24-months post-surgery
  Soft tissue retention will be evaluated utilising serial MRI imaging with assessment of soft tissue volume using a standardised segmentation protocol by a senior radiologist. Imaging will be taken at regular intervals in conjunction with clinical visits as defined by the protocol.
Preservation of pre-operative functional status | Assessed at 12-months post-surgery
  All patients prospectively enrolled in the trial will undergo pre-operative exercise tolerance testing to confirm their suitability for the trial. This is a standard test that each patient with Pectus Excavatum undergoes before any surgical operation. This will be repeated after complete recover from the operation (after 12 months) to evaluate whether the intervention has affected the patient's functional status. Standard cardiopulmonary exercise testing (CPET) protocol will be applied and validated by a physician.
Change in pain assessments from baseline to the end of study visit | Assessed at 1-month post surgery
  Pain will be assessed with the numerical pain rating system from 0 (no pain at all) to 10 (worst imaginable pain)
Change in wound healing from the time of surgery to the end of study visit | Assessed at 1-month post surgery
  Wound status will be assessed with the Holger Classification for wounds
Change in patient quality of life as assessed by Quality of Life (QoL) questionnaires from baseline to the end of study visit | Assessed at 3, 6, 12 and 24 month - clinical review
  The validated Italian translation of the 36-item Short Form Quality of Life (SF-36) questionnaire, a patient-reported survey of patient health, will be used to assess patient reported functional outcomes from the intervention. It consists of eight scaled scores (physical functioning, limitations due to physical health, limitations due to emotional problems, energy and fatigue, social role functioning, emotional well-being, bodily pain, general health perceptions), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100: the lower the score the more disability, the higher the score the less disability (a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability). The SF-36 questionnaire will be administered pre-operation and post-operation.

OTHER OUTCOMES:
Observational assessment of health economic measures from the time of surgery to the end of study visit | Assessed at 24 post-surgery months
  This will be assessed as a composite measure of:
  * Length of admission (measured in days), Infrastructure costs (measured in euro) and Operative time (measured in minutes) which will be monitored throughout the trial to provide a guide for optimisation of current protocols and potential translation into use of PCL scaffolds for reconstruction in broader clinical settings.
  * If patients undergo subsequent fat grafting, core biopsy samples will be taken in order to histologically evaluate the scaffold content. Specific stains will be used to assess tissue morphology, angiogenesis and immune activity. These can be correlated with medical imaging, as well as previous data gained from pre-clinical animal models.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Facchini, Dr, Principal Investigator — Unit of Paediatric Surgery and Burn Center - Meyer Children's Hospital
Locations (1):
- Meyer Children's Univeristy Hospital, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: No